CLINICAL TRIAL: NCT02624765
Title: FAST RCT: Prospective Randomized Clinical Trial of Fetal Atrial Flutter & Supraventricular Tachycardia Therapy
Brief Title: Prospective Randomized Clinical Trial of Fetal Atrial Flutter & Supraventricular Tachycardia Therapy (FAST RCT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Edgar Jaeggi (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Edgar Jaeggi, Edgar Jaeggi, MD FRCP (C), The Hospital for Sick Children
Organization: The Hospital for Sick Children (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000039945
Record Dates: First submitted 2015-11-30; First posted 2015-12-08 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Fetal Atrial Flutter Without Hydrops; Fetal Supraventricular Tachycardia Without Hydrops; Fetal Supraventricular Tachycardia With Hydrops
Keywords: RCT A: Fetal Atrial Flutter without Hydrops; RCT B: Fetal Supraventricular Tachycardia without Hydrops; RCT C: Fetal Supraventricular Tachycardia with Hydrops
MeSH Terms: interventions — Digoxin; Sotalol; Flecainide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- RCT A (1st arm): AF without hydrops (Active Comparator): Atrial Flutter (AF) without hydrops: Treatment with Digoxin as monotherapy.
  Interventions: Drug: Digoxin (monotherapy)
- RCT A (2nd arm): AF without hydrops (Active Comparator): Atrial Flutter (AF) without hydrops: Treatment with Sotalol as monotherapy.
  Interventions: Drug: Sotalol (monotherapy)
- RCT B (1st arm): SVT without hydrops (Active Comparator): Supraventricular Tachycardia (SVT) without hydrops: Treatment with Digoxin as monotherapy.
  Interventions: Drug: Digoxin (monotherapy)
- RCT B (2nd arm): SVT without hydrops (Active Comparator): Supraventricular Tachycardia (SVT) without hydrops: Treatment with Flecainide as monotherapy.
  Interventions: Drug: Flecainide (monotherapy)
- RCT C (1st arm): SVT with hydrops (Active Comparator): Supraventricular Tachycardia (SVT) with hydrops: Treatment with Digoxin and Sotalol.
  Interventions: Drug: Digoxin (dual therapy); Drug: Sotalol (dual therapy)
- RCT C (2nd arm): SVT with hydrops (Active Comparator): Supraventricular Tachycardia (SVT) with hydrops: Treatment with Digoxin and Flecainide.
  Interventions: Drug: Digoxin (dual therapy); Drug: Flecainide (dual therapy)

INTERVENTIONS:
Drug: Digoxin (monotherapy) — Oral or IV loading dose: 0.5 mg q 12 h (total 4 doses over 48 hours) followed by Oral maintenance dose: 0.25 mg-1mg/day
  Arms: RCT A (1st arm): AF without hydrops; RCT B (1st arm): SVT without hydrops
Drug: Sotalol (monotherapy) — Oral dose: 80 mg TID or 120 mg BID (240 mg/day)
  Arms: RCT A (2nd arm): AF without hydrops
Drug: Flecainide (monotherapy) — Oral dose: 100 mg TID (300 mg/day)
  Arms: RCT B (2nd arm): SVT without hydrops
Drug: Digoxin (dual therapy) — Oral or IV loading dose: 0.5 mg q 8 h (total 4 doses over 32 hours) followed by oral maintenance dose: 0.25 mg-1mg/day
  Arms: RCT C (1st arm): SVT with hydrops; RCT C (2nd arm): SVT with hydrops
Drug: Sotalol (dual therapy) — Oral dose: 160 mg BID (320 mg/day)
  Arms: RCT C (1st arm): SVT with hydrops
Drug: Flecainide (dual therapy) — Oral dose:100 mg TID (300 mg/day)
  Arms: RCT C (2nd arm): SVT with hydrops

SUMMARY:
The Fetal Atrial Flutter and Supraventricular Tachycardia (FAST) Therapy Trial is a prospective multi-center trial that examines the efficacy and safety of standard prenatal antiarrhythmic treatment. Study components of FAST include three prospective sub-studies to determine the efficacy and safety of commonly used transplacental drug regimens in suppressing fetal AF without hydrops (Randomized Clinical Trial (RCT) A), SVT without hydrops (RCT B), and SVT with hydrops (RCT C). All RCTs are open label phase III trials of standard 1st line therapy, which either is started as monotherapy (no hydrops) or as dual therapy (hydrops).

DETAILED DESCRIPTION:
Few studies are specifically designed to address health concerns relevant during pregnancy. The consequence is a lack of evidence on best clinical practice. This includes mothers and their babies when pregnancy is complicated by an abnormally fast heart rate up to 300 beats per minute due to supraventricular tachyarrhythmia (SVA) in the unborn baby (fetus). Although fetal SVA, including atrial flutter (AF) and other forms of supraventricular tachycardia (SVT), is the most common cause of intended in-utero fetal therapy, none of the medication used to date has been evaluated for their effects on the mother and her baby in a randomized controlled trial (RCT). As a consequence, physicians need to make decisions about the management of such pregnancies without any evidence from controlled trials on drug efficacy and safety and no consensus among specialists for the optimal management. The Fetal Atrial Flutter and Supraventricular Tachycardia (FAST) Therapy Trial is a prospective multi-center trial that addresses this knowledge gap to guide future fetal SVA therapy to the best of care. Study components of FAST include three prospective sub-studies to determine the efficacy and safety of commonly used transplacental drug regimens in suppressing fetal AF without hydrops (RCT A), SVT without hydrops (RCT B), and SVT with hydrops (RCT C). All RCTs are open label phase III trials of standard 1st line therapy, which either is started as monotherapy (no hydrops) or as dual therapy (hydrops). The primary study aim is the probability of a normal pregnancy outcome after treatment start with Digoxin or Sotalol (AF without hydrops); Digoxin or Flecainide (SVT without hydrops); and Digoxin plus Sotalol or Digoxin plus Flecainide (SVT with hydrops).

ELIGIBILITY:
Inclusion Criteria:

1. Mother has provided written informed consent to participate
2. Either fetal AF without hydrops, SVT without hydrops or SVT with hydrops
3. Tachyarrhythmia that is significant enough to justify immediate transplacental pharmacological treatment:

   * Tachycardia ≥ 180 bpm during at least 10% of observation time of 30 minutes or longer
   * Tachycardia ≥ 170 bpm during +100% of time (≤ 30 0/7 weeks of gestation)
   * Tachycardia ≥ 280 bpm (irrespective of SVA duration)
   * SVT with fetal hydrops (irrespective of duration)
4. Gestational age > 12 0/7 weeks and <36 0/7 weeks at time of enrollment
5. Untreated tachycardia at time of enrollment
6. Singleton Pregnancy
7. Healthy mother with ± normal pre-treatment cardiovascular findings:

   * ECG without significant abnormalities (sinus rhythm; QTc ≤ 0.47; PR ≤ 0.2 sec; QRS: ≤ 0.12 sec; isolated PACs or PVCs or isolated complete right bundle branch block allowed)
   * Resting heart rate ≥ 50 bpm
   * Systolic BP ≥ 85 bpm

Exclusion Criteria:

1. AF with hydrops (eligible for FAST Registry only)
2. Any maternal-fetal conditions associated with high odds of premature delivery or death other than tachycardia (e.g. severe IUGR; premature rupture of membrane; life-threatening maternal disease (incl. pre-eclampsia; HELLP syndrome); severe congenital fetal abnormalities (T 13 or 18; surgery or death expected < 1 month)
3. History of significant maternal heart condition (open heart surgery; sick sinus syndrome; channelopathy (long QT, Brugada syndrome); ventricular tachycardia; WPW syndrome; high-degree heart block; cardiomyopathy)
4. Relevant preexisting maternal obstructive airway disease including asthma
5. Current therapy with the following medications:

   * Antiarrhythmic drugs
   * Pentamidine
6. Maternal serum potassium level <3.3 mmol/L / <3.3 mEq/L (at start of treatment)
7. Maternal ionized serum calcium level of <1 mmol/L / <4 mg/dL) or total serum calcium level <2 mmol/L / <8mg/dL (at start of treatment)
8. Maternal serum creatinine level > 97.2 µmol/L (>1.1 mg/dl)

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Proportion of live-born children with a delivery at term and a normal cardiac rhythm | Term: 37 0/7 to 41 6/7 weeks
  Term delivery (≥37 0/7 weeks gestation) with a normal cardiac rhythm (ECG).

SECONDARY OUTCOMES:
Proportion of patients with cardioversion over time | From date of randomization until the date of first documented cardioversion or until the date of delivery/fetal death without cardioversion, whichever comes first, assessed up to 30 gestational weeks
  Number of participants with persistent tachycardia compared to number of participants with cardioversion to a normal rhythm over time
Proportion of participants with treatment failure | From date of randomization until the date of first documented fetal cardioversion or until the date of treatment failure, whichever comes first, assessed up to 30 gestational weeks
  Number of participants with treatment failure compared to number of participants with successful treatment. Treatment failure is defined as one of the following: 1) cross-over to another drug; 2) SVT/AF that persists to birth; 3) preterm birth; 4) death.
Proportion of participants with arrhythmia-related death | From date of randomization to 30 days of life
  Number of participants with arrhythmia-related death compared to other outcomes
Average gestational age at birth | At birth
  Mean of the gestational age at birth
Birth weight z-scores | At birth
  A birth weight z-score compares a child's birth weight to the weight of a child of the same length/height and gender to classify nutritional status
Total days of treatment related maternal and neonatal hospitalizations | From date of randomization to 30 days of life
  Average days of maternal and neonatal hospitalization related to SVA therapy
Maternal prevalence of adverse events and outcome | From date of randomization to 30 days of life
  Maternal prevalence of pregnancy/treatment-related AEs and outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Jaeggi, MD, Principal Investigator — The Hospital for Sick Children, Toronto
Locations (22):
- United States (12):
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's National Health System, Washington D.C., District of Columbia
  - Morgan Stanley Children's Hospital of New York-Presbyterian, New York, New York
  - Cohen Children's Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Pediatrix Medical Services, Inc,, Austin, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - West Virginia University Research Corporation, Morgantown, West Virginia
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- The Royal Women's Hospital, Melbourne, Victoria, Australia
- Canada (5):
  - University of Alberta/WCCHN, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Mount Sinai Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine Hospital, Montreal, Quebec
- UKB Universitätsklinikum BONN, Bonn, Germany
- Netherlands (2):
  - Academic Medical Center - AMC, Amsterdam
  - Leiden University Medical Center - LUMC, Leiden
- St George's University Hospital Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not planned

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-07): https://cdn.clinicaltrials.gov/large-docs/65/NCT02624765/Prot_SAP_000.pdf